CLINICAL TRIAL: NCT03977168
Title: A Prospective Study of Early Mechanical Stabilization and Bleeding in Disruption of the Pelvic Ring
Acronym: EMS-BIND
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: W81XWH-16-2-0060-EMS-BIND
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures | interventions — cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Application of circumferential pelvic compression (CPC) device — Application of circumferential pelvic compression (CPC) device used at any time within 24 hours of injury

SUMMARY:
The objective of this study is to evaluate the effect of earlier placement of Circumferential Pelvic Compression (CPC) on resuscitative measures required for life-threatening pelvic ring injuries and to guide the development of future efficacy trials of three advanced resuscitation techniques (surgical pelvic packing, angioembolization, REBOA).

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 18 and 64 years, inclusive;
* Severe blunt or blast traumatic injury;
* Young-Burgess APC-2 and 3, LC-3, vertical shear, and combined mechanism of injury (CMI) (Tile B and C patterns; OTA codes 61-B and 61-C);
* Circumferential pelvic compression (CPC) device used at any time within 24 hours of injury.
* Patient must speak either English or Spanish

Exclusion Criteria:

* Arrival to hospital of definitive care more than 6 hours after injury;
* Ballistic pelvic injury, other than from a blast mechanism;
* Time of CPC placement not recorded;
* Time of injury and time of EMS dispatch unknown;
* Use of medical anti-shock trousers (MAST);
* Confirmed dead on arrival to hospital

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with severe pelvic ring disruptions
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Blood products | 24 hours
  We will document the volume of any blood products given within the first 24 hours following injury
Pelvic stabilization and resuscitative techniques | 24 hours
  We will document any techniques used to stabilize and/or resuscitate the pelvic injury within the first 24 hours

SECONDARY OUTCOMES:
Blood loss | 24 hours
  Total blood volume loss will be calculated within the first 24 hours following injury
Ventilator days | 24 hours
  Number of days that patient spends on a ventilator will be documented
ICU days | 24 hours
  Number of days spent in the ICU will be documented
Length of hospital stay | 24 hours
  Number of days spent in the hospital will be documented
GCS (Glascow Coma Score) | 24 hours
  The GCS is a neurological scale to assess for brain injury. The score is composed of three parts: eyes, verbal and motor. Each component has a different scale. Eyes (1-4), verbal (1-5) and motor (1-6). The sum of all three components result in the overall GCS score (3-15). The higher the score, the less likelihood of brain injury

OTHER OUTCOMES:
Mortality | 1 month
  Any deaths that occur between index hospitalization and 30 days post-injury will be documented

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Methodist Hospital, Indianapolis, Indiana
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center - Houston, Houston, Texas
  - San Antonio Military Medical Center (SAMMC), San Antonio, Texas
  - University of Washington/Harborview Medical Center, Seattle, Washington